CLINICAL TRIAL: NCT07084727
Title: Retinal Biomarkers as a Tool for Early Detection of Endothelial Dysfunction in Women With Preeclampsia
Brief Title: Identifying Biomarkers for Endothelial Dysfunction in Women With Preeclampsia
Acronym: DAISY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 7765
Record Dates: First submitted 2025-07-01; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Endothelial Function (FMD); Preeclampsia; Retinal Vessels
MeSH Terms: conditions — Pre-Eclampsia | interventions — Vascular Stiffness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional group (Other): All patients in this study will undergo all vascular assessments including pulse wave velocity, pulse wave analysis, flow-mediated dilation, fundus photography and dynamic retinal vessel analysis.
  Interventions: Other: Arterial stiffness; Other: Flow-meditad dilatation; Other: Dynamic retinal vessel analyzer

INTERVENTIONS:
Other: Arterial stiffness — Non-invasive test. A blood pressure cuff and tonometer (a type of pen placed on the neck) are used to measure the speed at which a pressure wave propagates from one place to another.
  Every time the heart contracts, a pressure wave is generated that propagates from the heart to the blood vessels at a certain speed. The stiffer the blood vessels, the faster the wave propagates.
Other: Flow-meditad dilatation — This study measures the capacity with which blood vessels expand when we briefly cut off blood flow. The endothelium, the inner layer of blood vessels, regulates this expansion. By ultrasound, we measure the difference in diameter of the elbow artery. To cut off the blood flow, we clamp the forearm with a blood pressure cuff for 5 minutes.
  When the blood pressure cuff is released, it triggers increased blood flow in the arm, causing the blood vessels to expand. We record this expansion using the above techniques.
Other: Dynamic retinal vessel analyzer — Eye imaging measures the capacity with which your blood vessels in the retina can expand in response to a flicker light stimulation.

SUMMARY:
Every pregnancy has a major impact on a woman's heart and blood vessels due to changes required by the body to maintain proper blood flow between mother and foetus. When the placenta does not work properly, preeclampsia can occur. An important first symptom is high blood pressure. Women who have experienced preeclampsia are at higher risk of developing blood pressure and heart problems later on. Therefore, it is very important to detect changes in the blood vessel system so that they can be treated promptly and correctly. We aim to do this by using a new, non-invasive eye test that examines the blood vessels of the retina.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old
* willing to undergo vascular assessments
* informed consent signed

Exclusion Criteria:

* Unwilling to provide informed consent
* Open-angle glaucoma
* Epilepsia
* (gestational) Diabetes
* Multiple pregnancies
* Fetal malformations
* Hypercholesterolemia
* Kidney disease
* Auto-immune disorders
* Connective tissue diseases

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-11-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Retinal biomarkers | Baseline
  Early (retinal) biomarkers for cardiovascular risk in patients with preeclampsia, assessed by DVA.

CONTACTS AND LOCATIONS:
Locations (1):
- Antwerp University Hospital, Edegem, Antwerp, Belgium